CLINICAL TRIAL: NCT03313674
Title: Seasonal Affective Disorder: Exploratory Investigation of Seasonal Variations in Brain Structure and Connectivity as a Predictor for Depressive Severity
Brief Title: Investigation of Seasonal Variations of Brain Structure and Connectivity in SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Neurosurgeon, Scientist, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 281-2017
Record Dates: First submitted 2017-10-10; First posted 2017-10-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Seasonal Affective Disorder; Major Depressive Disorder; Neuroimaging
MeSH Terms: conditions — Seasonal Affective Disorder; Depressive Disorder, Major | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seasonal Affective Disorder (Experimental): The primary objective is to use neuroimaging paradigms to identify perturbations in neural circuits of SAD patients when they are clinically depressed in the winter, after bright light therapy treatment, and when they are healthy in the summer
  Interventions: Device: Bright Light Therapy
- Major Depressive Disorder (No Intervention): SAD patients will be compared to unipolar depressed patient cohort, who will be imaged in the winter and the summer.
- Healthy Controls (No Intervention): SAD patients will be compared to healthy controls, who will be imaged in the winter and the summer.

INTERVENTIONS:
Device: Bright Light Therapy — Light box that emits light at 10,000 lux or higher and has been demonstrated to regulate circadian rhythm that is aberrant in the SAD population
  Arms: Seasonal Affective Disorder

SUMMARY:
Seasonal Affective Disorder (SAD) is a subtype of Major Depressive Disorder, characterized by a recurrent temporal relationship between the season of year, the onset and the remission of a major depressive episode. Estimates of the annual prevalence state that 1-6% of the population will develop SAD with the larger prevalences found at greater extremes in latitude. SAD is most likely triggered by the shortening photoperiod experienced in the winter months leading to a deterioration of mood. Recent cross-sectional neuroimaging studies have found cellular and neurotransmitter changes in response to seasonality, ultimately having an impact on the affect of patients. Conversly, this study aims to investigate the changes in neurocircuitry related to depression and euthymic states. Patients with SAD offer a unique ability to study these changes since they have predictable triggers for the onset of depression (i.e. the winter months) and remission (i.e. the summer months).

ELIGIBILITY:
Inclusion Criteria for SAD Cohort

1. Male or female between the ages of 18 to 65 years, inclusive
2. Patients who are able and willing to give consent and able to attend study visits
3. Agreement to use light therapy for four weeks
4. DSM-V diagnosis of seasonal affective disorder, at least 2 year history of the illness with a Structured Interview Guide for the Hamilton Depression Rating Scale-SAD version (SIGH-SAD) score ≥ 25 at screening

Exclusion Criteria for SAD Cohort

1. Current alcohol and/or substance use disorder
2. Use of cigarettes
3. Past or present psychiatric disorders (axis I and II) other than SAD
4. Taken medications approved and/or employed off-label for depression
5. Previous use of light therapy
6. Use of photosensitive medications
7. Montreal Cognitive Assessment score < 24
8. Patients with standard contraindications for MR imaging. For example, non-MRI compatible metallic implants including cardiac pacemaker, size limitations etc.
9. Known intolerance or allergies to MRI contrast agent (Gadolinium or Magnevist) including advanced kidney disease
10. Severely impaired renal function (estimated glomerular filtration rate <30ml/min/1.73m2)
11. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
12. Pregnant and/or breastfeeding
13. Travelled to another a more southern latitude within 6 months of scan
14. Night shift workers
15. Are participating or have participated in clinical trial or research study in the last 30 days
16. Unable to communicate with investigator and/or staff
17. Diagnosis of a reading disability, dyslexia or significant learning disorder

Inclusion Criteria for Unipolar Depression Cohort contraindications

1. Male or female between the ages of 18 to 65 years, inclusive
2. Patients who are able and willing to give consent and able to attend study visits
3. DSM-V diagnosis of major depressive disorder, with a Hamilton Depression Rating Scale score ≥ 22 at screening

Exclusion Criteria for Unipolar Depression Cohort

1. Current alcohol and/or substance use disorder
2. Past or present psychiatric disorders (axis I and II) other than SAD
3. Montreal Cognitive Assessment score < 24
4. Patients with standard contraindications for MR imaging. For example, non-MRI compatible metallic implants including cardiac pacemaker, size limitations etc.
5. Known intolerance or allergies to MRI contrast agent (Gadolinium or Magnevist) including advanced kidney disease
6. Severely impaired renal function (estimated glomerular filtration rate <30ml/min/1.73m2)
7. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
8. Pregnant and/or breastfeeding
9. Are participating or have participated in clinical trial or research study in the last 30 days
10. Unable to communicate with investigator and/or staff
11. Diagnosis of a reading disability, dyslexia or significant learning disorder

Inclusion Criteria for Healthy Controls

1. Male or female between the ages of 18 to 65 years, inclusive
2. Patients who are able and willing to give consent and able to attend study visits
3. No current or past history of mental disorder
4. No unstable medical disorders

Exclusion Criteria for Healthy Controls

1. Use of any medication for a general medical disorder and/or condition that, in the opinion of the investigator, may affect neural structure
2. Alcohol or drug-use within 24 hours of MRI
3. Pregnant and/or breastfeeding
4. Montreal Cognitive Assessment score < 24
5. Patients with standard contraindications for MR imaging. For example, non-MRI compatible metallic implants including cardiac pacemaker, size limitations etc.
6. Known intolerance or allergies to MRI contrast agent (Gadolinium or Magnevist)
7. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
8. Are participating or have participated in clinical trial or research study in the last 30 days
9. Unable to communicate with investigator and/or staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Changes in neural function | 12 months
  Functional MRI Scan
Changes in connectivity | 12 months
  Diffusion Tensor Imaging Scan

SECONDARY OUTCOMES:
Executive Function | 12 months
  Trail Makers Test B will be used to measure executive function. Test is scored based on time to complete.Average time is 75 seconds, deficient time is >273 seconds
Concentration | 12 months
  Digit Symbol Substitute Test will be used to measure concentration. Survey score is determined by the number of correct and incorrect responses
Memory | 12 months
  California Verbal Learning Test. Score is conducted based on a propriety software based on the number of correctly recalled words after a list is administrated.
Blood Serum Metabolomic seasonal variation | 12 months
  Blood will be drawn to assess different serum metabolites depending on the season. One blood draw will be taken in Winter, one in the summer. Over 3300 metabolites will be acquired from a single sample.
Depressive severity measured through the • Structured Interview Guide for the Hamilton Depression Rating Scale-SAD version | 12 months
  Sigh-SAD measures Depressive Severity specifically in SAD patients. It contains 29 items, with the total score ranging from 0 to 29. Higher values in the scale indicate worse depression severity.
  Of the 29 items, 21 question (adapted from the Hamilton Depression scale) are used to determine typical depression severity, with an additional eight items for the "atypical" symptoms which are presented in seasonal affective disorder. The final score is summed, with equal weighting, to give the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No